CLINICAL TRIAL: NCT02061371
Title: VIRTUAL THERAPY IN REHABILITATION SPASTIC HEMIPARESIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 20749113.5.0000.5503
Record Dates: First submitted 2014-02-07; First posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-01

CONDITIONS: Stroke
Keywords: stroke; spasticity; physiotherapy; virtual reality
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- virtual therapy (Experimental): Group 1 (G1) included 20 patients who will carry out the virtual therapy.
  Interventions: Other: virtual therapy
- conventional physiotherapy (Experimental): Group 2 (G2) included 20 patients who hold conventional physiotherapy.
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Other: virtual therapy
  Arms: virtual therapy
Other: conventional physiotherapy
  Arms: conventional physiotherapy

SUMMARY:
Evaluate the effectiveness of virtual therapy and conventional physiotherapy in spastic muscles of patients with sequelae of stroke.

DETAILED DESCRIPTION:
Considered the second most frequent cause of death worldwide , the stroke is also responsible for the largest number of functional disability in individuals. The socio - economic hardship that many patients face to perform a program of intensive rehabilitation sensorimotor, has led to functional limitations in many cases , promote irreversible consequences. Spasticity in the upper and lower limb after stroke results in loss of function and mobility being the key therapeutic approaches in order to restore its function. Currently, the Virtual therapy has been used in physical therapy, demonstrating safety, feasibility and potential to facilitate the effective rehabilitation treatment, promoting motor recovery. The objective of this study is to analyze and compare the effectiveness of virtual therapy and conventional physiotherapy in paretic upper and lower limbs of patients with sensory motor deficit after stroke. Virtual therapy will be based on a custom application using virtual reality projection, and conventional treatment will be based on cinesiotherapy for members upper and lower paretic. The evaluation will be performed by biomedical instrumentation using dynamometry, electromyography and analysis from functional movement. Statistical differences are based on t test with significance level of p 0 , 05 . As a result expected - scientifically proven the effectiveness of this new form of treatment aimed at improving quality of life and functional independence of patients with neurological sequel.

ELIGIBILITY:
Inclusion Criteria:

* Medical referral for physiotherapy;
* Maximum grade 2 spasticity in the upper and lower limbs according to the Modified Ashworth Scale;
* Total passive range of elbow joint and knee to the movement of flexion and extension;
* Independent ambulation, with or without support;
* Cognitive preserved, being able to respond to the command of the examiner;
* Least 6 months of injury;

Exclusion Criteria:

* Active infection, and rash at the site of application of NMES;
* Visual and hearing impairment;
* Joint stiffness and musculoskeletal injuries of the elbow and knee,
* Inability to interpret the therapeutic resources to be displayed;
* Presenting lesions in areas of Wernick and drill;
* Uncontrolled hypertension.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Espasticity | 4 months
  It is believed that this study achieves positive results regarding the adequacy of muscle tone associated with musculoskeletal better performance, so that the muscles normotônicos gain strength and overcome the resistance of the hypertonic muscles, improving range of motion and harmony of the affected limbs, leading the consequent improvement of balance and gait, after application of virtual therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Lersm, Ip&D, São José dos Campos, São Paulo, Brazil